CLINICAL TRIAL: NCT03632460
Title: Comparison of Epidural Dexmedetomidine and Dexamethasone as an Adjuvant to Ropivacaine on Postoperative Pain Level, Analgesic Consumption and Oxidative Stress in Thoracic Surgery
Brief Title: Dexmedetomidine and Dexamethasone as an Adjuvant to Ropivacaine in Thoracic Surgery
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University Hospital Dubrava (Other)
Responsible Party: Principal Investigator, Jasminka Persec, MD, PhD, Assist Prof MD PhD, University Hospital Dubrava
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: UHDubrava777
Record Dates: First submitted 2018-08-08; First posted 2018-08-15 (Actual); Last update posted 2018-08-15 (Actual); Status verified 2018-08

CONDITIONS: Pain, Postoperative; Oxidative Stress
MeSH Terms: conditions — Pain, Postoperative | interventions — Dexmedetomidine

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Dexmedetomidine (Active Comparator): 1 mcg/kg dexmedetomidine added to 8 ml 0.375% ropivacaine
  Interventions: Drug: Dexmedetomidine Injection [Precedex]
- Dexamethasone (Active Comparator): 8 mg dexamethasone added to 8 ml 0,375% ropivacaine
  Interventions: Drug: Dexmedetomidine Injection [Precedex]

INTERVENTIONS:
Drug: Dexmedetomidine Injection [Precedex] — epidural administration of dexmedetomidine added to ropivacaine

SUMMARY:
The aim of the study is to investigate the effect of preoperative epidural dexmedetomidine compared to dexamethasone on postoperative pain control, analgesic consumption and oxydative stress response in patients undergoing thoracic surgery

DETAILED DESCRIPTION:
The aim of the study is to investigate the effect of preoperative epidural dexmedetomidine compared to dexamethasone on postoperative pain control, analgesic consumption and oxydative stress response in patients undergoing thoracic surgery.

Investigation will include patients between 30-70 years undergoing thoracic surgery due to malignant process of lung or oesophagus.

Patients are divided in two groups: epidural administration of 0.375% ropivacaine with 1 mcg/kg dexmedetomidine (group 1) and epidural administration of 0.375% ropivacaine with 8 mg dexamethasone.

ELIGIBILITY:
Inclusion Criteria:

* patients undergoing thoracic surgery due to malignant process of lung or oesophagus ASA (American Society of Anesthesiologists) status I-III

Exclusion Criteria:

* neurological or psychiatric disease
* corticosteroid therapy
* anamnesis of myocardial infarct within last 6 months
* severe aortic stenosis
* kidney insufficiency
* liver insufficiency
* allergy
* coagulation disorders

Ages: 30 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2018-09-01 (Estimated); Primary Completion 2018-12-31 (Estimated); Study Completion 2019-05-01 (Estimated)

PRIMARY OUTCOMES:
Change in postoperative pain level using visual analogue scale | Before operation, 1 hour, 2 hour, 6 hour and 24 hour after operation
  Change in baseline postoperative pain level measured before operation, and then at 1h, 2h, 6h and 24h after operation using visual analogue scale. Visual analogue scale is numerical scale in range from 1-10, assessing pain level. Minimum score is 1, which represents- no pain to maximum score 10 which represents- the worst pain ever experienced.

SECONDARY OUTCOMES:
analgesic consumption | 24 hour
  analgesic consumption in time interval
oxydative stress level | 24 hour
  malonyldialdehyde, glutathion, catalase

CONTACTS AND LOCATIONS:
Overall Officials: Jasminka Persec, Assit Prof, Principal Investigator — University Hospital Dubrava; Andrej Sribar, MD, Study Chair — University Hospital Dubrava
Locations (1):
- Jasminka Persec, Zagreb, Croatia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Kim NY, Kwon TD, Bai SJ, Noh SH, Hong JH, Lee H, Lee KY. Effects of dexmedetomidine in combination with fentanyl-based intravenous patient-controlled analgesia on pain attenuation after open gastrectomy in comparison with conventional thoracic epidural and fentanyl-based intravenous patient-controlled analgesia. Int J Med Sci. 2017 Aug 18;14(10):951-960. doi: 10.7150/ijms.20347. eCollection 2017. PMID 28924366
- [Result] Hong JM, Kim KH, Lee HJ, Kwon JY, Kim HK, Kim HJ, Cho AR, Do WS, Kim HS. Epidural Dexamethasone Influences Postoperative Analgesia after Major Abdominal Surgery. Pain Physician. 2017 May;20(4):261-269. PMID 28535549
- [Result] Gallego-Ligorit L, Vives M, Valles-Torres J, Sanjuan-Villarreal TA, Pajares A, Iglesias M. Use of Dexmedetomidine in Cardiothoracic and Vascular Anesthesia. J Cardiothorac Vasc Anesth. 2018 Jun;32(3):1426-1438. doi: 10.1053/j.jvca.2017.11.044. Epub 2017 Dec 2. PMID 29325842